CLINICAL TRIAL: NCT02311621
Title: A Phase 1 Feasibility and Safety Study of Cellular Immunotherapy for Recurrent/Refractory Neuroblastoma Using Autologous T-cells Lentivirally Transduced to Express CD171-specific Chimeric Antigen Receptors
Brief Title: Engineered Neuroblastoma Cellular Immunotherapy (ENCIT)-01
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: The Evan Foundation (Other); Ben Towne Center for Childhood Cancer Research (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENCIT-01
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Neuroblastoma; Ganglioneuroblastoma
Keywords: CAR T cell; pediatric; young adults
MeSH Terms: conditions — Neuroblastoma; Ganglioneuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- A: 2nd Generation CE7R CAR T Cells (Experimental): Autologous CD4 and CD8 cells are lentivirally transduced to generate patient-derived CD171 specific CAR T cells also expressing an EGFRt.
  Patients will receive lymphodepletion chemotherapy prior to T cell infusion. CD171 specific CAR T cells will be administered approximately 2-3 days after lymphodepletion chemotherapy.
  Cells will be administered approximately 1:1 CD4 and CD8 cells with planned dose level evaluations of total T cell dose of 1x10^6 cells/kg, 5x10^6 cells/kg, 1x10^7 cells/kg, 5x10^7 cells/kg, and 1x10^8 cells/kg will be evaluated.
  Interventions: Biological: Patient Derived CD171 specific CAR T cells expressing EGFRt (2nd generation T cells)
- B: 3rd Generation CE7R CAR T Cells (Experimental): Autologous CD4 and CD8 cells are lentivirally transduced to generate patient-derived CD171 specific CAR T cells also expressing an EGFRt.
  Patients will receive lymphodepletion chemotherapy prior to T cell infusion. CD171 specific CAR T cells will be administered approximately 2-3 days after lymphodepletion chemotherapy.
  Cells will be administered approximately 1:1 CD4 and CD8 cells with planned dose level evaluations of total T cell dose of 1x10^6 cells/kg, 5x10^6 cells/kg, 1x10^7 cells/kg, 5x10^7 cells/kg, and 1x10^8 cells/kg will be evaluated.
  Interventions: Biological: Patient Derived CD171 specific CAR T cells expressing EGFRt (3rd generation T cells)
- C: Long Spacer 2nd Generation CE7R CAR T Cells (Experimental): Autologous CD4 and CD8 cells are lentivirally transduced to generate patient-derived CD171 specific CAR T cells also expressing an EGFRt.
  Patients will receive lymphodepletion chemotherapy prior to T cell infusion. CD171 specific CAR T cells will be administered approximately 2-3 days after lymphodepletion chemotherapy.
  Cells will be administered approximately 1:1 CD4 and CD8 cells with planned dose level evaluations of total T cell dose of 1x10^6 cells/kg, 5x10^6 cells/kg, 1x10^7 cells/kg, 5x10^7 cells/kg, and 1x10^8 cells/kg will be evaluated.
  Interventions: Biological: Patient Derived CD171 specific CAR T cells expressing EGFRt (long spacer 2nd generation T cells)

INTERVENTIONS:
Biological: Patient Derived CD171 specific CAR T cells expressing EGFRt (2nd generation T cells) — Intravenous infusion of autologous T cells transduced to express 4-1BB:zeta CD171CAR and EGFRt (2nd generation T cells)
  Arms: A: 2nd Generation CE7R CAR T Cells
Biological: Patient Derived CD171 specific CAR T cells expressing EGFRt (3rd generation T cells) — Intravenous infusion of autologous T cells transduced to express CD28:4-1BB:zeta CD171CAR and EGFRt
  Arms: B: 3rd Generation CE7R CAR T Cells
Biological: Patient Derived CD171 specific CAR T cells expressing EGFRt (long spacer 2nd generation T cells) — Intravenous infusion of autologous T cells transduced to express 4-1BB:zeta CD171CAR and EGFRt (long spacer 2nd generation T cells)
  Arms: C: Long Spacer 2nd Generation CE7R CAR T Cells

SUMMARY:
Patients with recurrent or refractory neuroblastoma are resistance to conventional chemotherapy. For this reason, the investigators are attempting to use T cells obtained directly from the patient, which can be genetically modified to express a chimeric antigen receptor (CAR). The CAR enables the T cell to recognize and kill the neuroblastoma cell through the recognition of CD171, a protein expressed of the surface of the neuroblastoma cell in patients with neuroblastoma. This is a phase 1 study designed to determine the maximum tolerated dose of the CAR+ T cells.

DETAILED DESCRIPTION:
Upon meeting the eligibility requirements and enrolling on study, subjects will undergo apheresis to obtain the T cells for the generation of the CD171 CAR+ T cells. The T cells are isolated from the apheresis product, the CD4 and CD8 T cells are then selected and grown separately, transduced with a lentivirus to express the CD171 CAR as well as a truncated EGFR that has no signaling capacity (noted EGFRt) and expanded in culture over a 4-6 week period. During the process of cell generation, subjects will continue to be cared for by their primary oncologist and may undergo additional treatment directed at neuroblastoma during this time.

After the CAR+ T cells have been generated, the subject undergoes a disease assessment and determination of necessary lymphodepletion therapy. A variety of lymphodepletion strategies are acceptable and determined on a case by case basis. At least 48 hours after the completion of lymphodepletion, the subject will receive and infusion of CAR+ T cells at an approximate 1:1 ratio of CD4 to CD8 CAR+ T cells.

Following treatment with the CAR+ T cells, subjects will be followed intensely for 6 weeks with serial blood testing and re-evaluation of disease status with MIBG scintigraphy, tumor imaging by MRI/CT and bone marrow aspirates. After 4-6 weeks, the subjects clinical care will be resumed by their primary oncologist, and it is possible that they would receive additional chemotherapy or investigational agents.

Some subjects will receive cetuximab for ablation of the genetically modified T cells. Criteria to receive cetuximab include acute toxicities that are life threatening, as well as studies indicating lymphoproliferative disorder arising from an infused genetically modified T cell.

Upon completion of the study, subjects will be followed bi-annually for 5 years, and then annually for 10 additional years with either a medical history, physical exam and blood tests or a phone call/questionnaire. This follow up will help to determine if the subject develops any long-term health problems related to the CAR+ T cells including a new cancer.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of NB or ganglioneuroblastoma either by histologic verification and/or demonstration of tumor cells in the bone marrow with increased catecholamine levels.
* Male or female subjects ≤ 26 years of age
* Diagnosis of high risk NB at initial diagnosis or if non-high risk at time of initial diagnosis must have had evidence of metastatic progression when > 18 months of age.
* Measurable or evaluable disease
* Lansky or Karnofsky performance status score of ≥ 50
* Life expectancy of ≥ 8 weeks.
* Recovered from significant acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to enrollment onto this study.
* ≥ 7 days since last chemotherapy or biologic therapy administration
* No systemic corticosteroids (unless physiologic replacement dosing) within 7 days of enrollment. Topical Administration (e.g. inhaled or dermatologic) is allowed.
* ≥ 3 half-lives or 30 days from time of last dose of anti-tumor directed antibody therapy, whichever is shorter from time of enrollment
* ≥ 6 weeks from myeloablative therapy and autologous stem cell transplant (timed from stem cell infusion). Patients who received stem cell infusion following non-myelo-ablative therapy are eligible once they meet all other eligibility requirements. Patient must NOT have received a prior allogeneic hematopoietic stem cell transplant.
* No prior genetically modified cell therapy that is still detectable.
* Must not be receiving external beam radiation therapy at the time of study enrollment. ≥ 12 weeks from prior I131 MIBG therapy.
* Adequate organ function
* Adequate laboratory values
* Negative HIV antigen and antibody, Hepatitis B surface antigen and Hepatitis C antibody within 3 months prior to enrollment. For patients with positive Hepatitis C Ab, negative PCR testing must be documented in order to be eligible.

Exclusion Criteria:

* History of relevant CNS pathology or current relevant CNS pathology (non-febrile seizure disorder requiring ongoing anti-epileptic medications, paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injuries, dementia, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder). Patients may have CNS intracranial tumor.
* Pregnant or breast-feeding
* Unable to tolerate apheresis procedure including placement of temporary apheresis catheter if necessary
* Presence of active malignancy other than NB
* Presence of known intracranial metastatic neuroblastoma. Skull based disease with soft tissue extension is allowed.
* Presence of active severe infection
* Presence of any concurrent medical condition that, in the opinion of the protocol PI or designee, would prevent the patient from undergoing protocol-based therapy.
* Presence of a primary immunodeficiency/bone marrow failure syndrome
* Receiving any other anti-cancer agents or radiotherapy at the time of study entry
* Unwilling or unable to provide consent/assent for participation in the study and 15-year follow-up

Ages: 18 Months to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2014-11-25 (Actual); Primary Completion 2023-11 (Actual); Study Completion 2038-11 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 28 days
  Patients will be evaluated through day 28 for occurrence of dose limiting toxicity

SECONDARY OUTCOMES:
Response (Tumor response will be evaluated by the revised International Neuroblastoma Response Criteria) | 42 days
  Tumor response will be evaluated by the revised International Neuroblastoma Response Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Albert, MD, Study Chair — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
Current plan will be to present as a combined data set once enrollment and assessments are complete. Individual data may be made available if clinically applicable based on extreme response or toxicity.